CLINICAL TRIAL: NCT02992704
Title: Randomised Control Study for Inactive Chronic Hepatitis B Patients With Low Viral Load, With Peg-Interferon (INACTIVE)
Brief Title: Peg-interferon for Inactive Chronic Hepatitis B Carriers
Acronym: INACTIVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seng Gee Lim (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Seng Gee Lim, Director of Hepatology, National University Health System, Singapore
Organization: National University Health System, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00205
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis, B Virus; Carrier of Viral Hepatitis Type B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Intervention Model Description: Three arm, parallel open label study
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG 24 weeks (Experimental): peginterferon alpha 2a 180mcg for 24 weeks
  Interventions: Drug: Peginterferon Alfa-2A
- PEG 48 weeks (Experimental): peginterferon alpha 2a 180mcg 48 weeks
  Interventions: Drug: Peginterferon Alfa-2A
- Control (No Intervention): No treatment for 72 weeks

INTERVENTIONS:
Drug: Peginterferon Alfa-2A — peginterferon alpha 2a 180mcg weekly for either 24 or 48 weeks
  Other Names: pegasys
  Arms: PEG 24 weeks; PEG 48 weeks

SUMMARY:
Chronic Hepatitis B carriers (normal LFTs and viral load < 2 x 10^4 IU/ml are not recommended to be treated by guidelines as they are at low risk for complications. However, it is unclear if treatment can enhance HBsAg loss which has been shown to be associated with significantly lower risk of complications compared to those without HBsAg loss. Consequently, this is a proof of concept study to determine the possibility of HBsAg loss in Chronic Hepatitis B carriers in a randomised open label clinical trial comparing no treatment to 24 weeks peg-interferon alpha 2a or 48 weeks peginterferon alpha 2a (randomised 1:1:1). The primary endpoint of HBsAg loss will be evaluated 24 weeks after the end of therapy for those on therapy and matched to an equivalent timepoint in the control arm. The sample size calculation is 30 patients in each arm for a 20% difference between any experimental arm and the control arm.

DETAILED DESCRIPTION:
1. Hypothesis: Chronic hepatitis B carriers (defined as HBeAg negative hepatitis B patients with HBV DNA <2x104 IU/mL, absence of cirrhosis and normal ALT) may experience higher rates of HBsAg seroclearance with pegylated interferon therapy.

2A. Primary Objective

* The proportion of subjects with HBsAg loss at Week 24 of followup after treatment with 24 or 48 weeks of pegylated interferon alpha 2a compared to no therapy.

  2B. Secondary Objective
* The proportion of subjects who experience HBsAg loss with 24 versus 48 weeks of pegylated interferon at the end of treatment, and at end of followup.
* The rate of quantitative HBsAg decline in relation to HBsAg loss
* The proportion of subjects with virological response (HBV DNA level <13.5IU/mL) at Weeks 12 and 24 of treatment, and week 24 of followup.

  2C Study population: 90 patient will be enrolled.

3.1 Inclusion Criteria

For entry into this study, the following inclusion criteria must be met:

* Males or females age 21-75 years old (inclusive)
* Treatment naïve
* Documented HBsAg or HBV DNA positive for ≥ 6 months.
* Documented HBeAg negative and anti-HBe positive
* ALT ≤1xULN
* quantitative HBsAg <1,000 IU/ml OR HBV DNA <2x104 IU/mL at screening
* Absence of cirrhosis documented by liver biopsy or transient elastography within 6 months (Fibroscan®; Fibrosis stage >2 (score ≥ 10Kpa) will not be eligible for this study.)
* Patient has agreed not to take any other investigational drug or systemic anti-viral, cytotoxic, corticosteroid, immunomodulatory agents or Chinese traditional remedies unless clinically indicated.
* Patient is able to give written consent prior to study start and to comply with the study requirements.
* Women of childbearing age must have a negative urine (ß-HCG) pregnancy test taken within 14 days of starting therapy

3.2 Exclusion Criteria

For entry into this study, the following exclusion criteria must not be met:

* Patients who are currently on treatment with nucleoside/nucleotide analogues or have been treated for Hepatitis B in the past
* Presence of cirrhosis documented by liver biopsy or transient elastography (score ≥ 10kpa)
* Active Co-infection with HIV antibody, HCV antibody or HDV antibody positivity.
* Evidence of decompensated liver disease defined as a direct (conjugated) bilirubin >1.2x upper limit of normal (ULN), prothrombin time (PT) >1.5xULN , serum bilirubin <35g/L, or prior history of clinical hepatic decompensation as illustrated by presence of (eg. ascites, encephalopathy, variceal haemorrhage)
* Evidence of hepatocellular carcinoma
* Absolute neutrophil count <1.5x10^9/L or Hemoglobin <12 g/L for men or <11 g/L for women, or platelet count < 90x10^9/L
* History of depression or psychiatric disease
* Uncontrolled thyroid disease defined as thyroid-stimulating hormone (TSH) >1.2 ULN or 0.8xLLN or thyroid dysfunction
* Any immunomodulators, systemic cytotoxic agents, or systemic cortiosteriods within 6 months before trial entry
* Significant renal, cardiovascular, pulmonary, neurological, autoimmune disease or bone disease (e.g., osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochrondroses, multiple bone fractures)
* Malignant disease within 5 years of trial entry
* Women who are pregnant and who are not practicing adequate birth control measures, (defined as two methods of birth control with at least one barrier method) or who are lactating.

4.1 Study Treatment

Product, Dose, and Mode of Administration:

Peginterferon α-2a (PEG), 180mcg, will be administered weekly by subcutaneous injection for the specified period of time (see Study Design, Arms B and C). Pegasys® (Roche Pharmaceuticals).

Reference Therapy, Dose, and Mode of Administration:

Peginterferon α-2a (PEG), 180mcg subcutaneous injection once weekly

4.2 Overview The study will be conducted as a computer randomised clinical trial with concealment of allocation. Patients fulfilling inclusion and exclusion criteria will be randomised after completing screening. Patients will be randomly allocated to three parallel arms: no therapy, 24 weeks peg-interferon alpha 2a, and 48 weeks interferon alpha 2a. Patients will be monitored 4 weekly initial then 12 weekly till end of therapy, then for an additional 24 weeks after completing therapy. Patients on no therapy will be monitored for 72 weeks.

4.3 Endpoints/efficacy assessements Primary: HBsAg loss at end of followup for interferon arms compared to no therapy

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* Documented HBsAg or HBV DNA positive for ≥ 6 months.
* Documented HBeAg negative and anti-HBe positive
* ALT ≤1xULN
* quantitative HBsAg <1,000 IU/ml
* HBV DNA <2x104 IU/mL at screening
* Absence of cirrhosis documented by liver biopsy or transient elastography within 6 months (Fibroscan®; Fibrosis stage >2 (score ≥ 10Kpa) will not be eligible for this study.)
* Patient has agreed not to take any other investigational drug or systemic anti-viral, cytotoxic, corticosteroid, immunomodulatory agents or Chinese traditional remedies unless clinically indicated.
* Patient is able to give written consent prior to study start and to comply with the study requirements.
* Women of childbearing age must have a negative urine (ß-HCG) pregnancy test taken within 14 days of starting therapy

Exclusion Criteria:

* Patients who are currently on treatment with nucleoside/nucleotide analogues or have been treated for Hepatitis B in the past
* Presence of cirrhosis documented by liver biopsy or transient elastography (score ≥ 10kpa)
* Active Co-infection with HIV antibody, HCV antibody or HDV antibody positivity.
* Evidence of decompensated liver disease defined as a direct (conjugated) bilirubin >1.2x upper limit of normal (ULN), prothrombin time (PT) >1.5xULN , serum bilirubin <35g/L, or prior history of clinical hepatic decompensation as illustrated by presence of (eg. ascites, encephalopathy, variceal haemorrhage)
* Evidence of hepatocellular carcinoma
* Absolute neutrophil count <1.5x10^9/L or Hemoglobin <12 g/L for men or <11 g/L for women, or platelet count < 90x10^9/L
* History of depression or psychiatric disease
* Uncontrolled thyroid disease defined as thyroid-stimulating hormone (TSH) >1.2 ULN or 0.8xLLN or thyroid dysfunction
* Any immunomodulators, systemic cytotoxic agents, or systemic cortiosteriods within 6 months before trial entry
* Significant renal, cardiovascular, pulmonary, neurological, autoimmune disease or bone disease (e.g., osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochrondroses, multiple bone fractures)
* Malignant disease within 5 years of trial entry
* Women who are pregnant and who are not practicing adequate birth control measures, (defined as two methods of birth control with at least one barrier method) or who are lactating.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
HBsAg loss | 24 weeks after end of therapy
  Qualitative HBsAg assay reads "non-detectable"

SECONDARY OUTCOMES:
HBsAg loss | At the end of 24 and 48 weeks of peginterferon therapy
  Qualitative HBsAg assay reads "non-detectable"
Decline in quantitative HBsAg level | At week 24, 48 and 24 weeks after completion of therapy
  Based on quantitative HBsAg assay
proportion of patients with undetectable HBV DNA | At week 24, 48 of therapy, and 24 weeks after end of therapy
  HBV DNA assay<13.5 IU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Seng Gee Lim, MBBS, FRACP, FRCP, MD, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No